CLINICAL TRIAL: NCT07033364
Title: Changes in Functional Liver Tissue After Liver Metastasis Irradiation: Pilot Study of Functional Imaging Before and After Stereotactic Body Radiotherapy
Brief Title: Functional Liver After SBRT
Acronym: FAFOR
Status: Recruiting | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: N25FAF
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Liver Metastases
Keywords: liver function test; functional liver imaging; hepatobiliary scintigraphy; dose effect relationship; radiotherapy; SBRT; nuclear medicine; liver function; HEBIS; HIDA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with liver metastases: Ten to fifteen patients with a single liver metastasis who will be treated with SBRT, will be included to assess functional imaging using HEBIS before and 3-4 months after their treatment (SBRT). Patients are included in a single institute in the Netherlands.
  Interventions: Other: Functional liver imaging using hepatobiliary scintigraphy (HEBIS)

INTERVENTIONS:
Other: Functional liver imaging using hepatobiliary scintigraphy (HEBIS) — The Hepatobiliary scintigraphy (HEBIS) or HIDA scan is a nuclear imaging technique that uses [99mTc]Tc-mebrofenin, a iminodiacetic acid (IDA) agent, which is a lidocaine analogue that is taken up by hepatocytes and is eliminated in the biliary tract (Arntz, 2023). This functional liver scan quantitatively assesses liver function of which the potential will be tested to measure liver function before and after radiotherapy.

SUMMARY:
In this study, the investigators aim to determine the dose-effect relationship between radiation dose and liver function by performing a hepatobiliary scintigraphy (HEBIS) before and after stereotactic body radiotherapy (SBRT) for patients with liver metastases. HEBIS is a nuclear imaging technique to quantitatively assess liver function. It better predicts the risk of postsurgical liver failure compared to volumetry alone. To prevent liver failure after SBRT, current clinical dose constraints require that ≥ 700 ml of normal liver should receive less than 15 Gy in 3 fractions. The exact local dose-effect relation is however unknown. Doses below 15 Gy are still damaging, while liver tissue receiving doses above 15 Gy will retain some function. By associating the 3D radiation dose distribution with the HEBIS scan, the investigators can evaluate the impact of radiation dose on liver function for different dose levels in liver (sub)volumes. This analysis will refine existing dose-effect relationships, enabling more tailored treatment of liver metastases in the future. Ten to fifteen patients will be included to assess functional liver imaging using HEBIS before their treatment and 3 to 4 months after their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated for a liver metastasis with SBRT with treatment prescription of 3 x 20 Gy
* Able to provide informed consent prior to any study specific procedure

Exclusion Criteria:

* WHO > 2
* Pregnancy
* Prior radiation therapy of the liver
* Lactation, unable to substitute for 24 hours
* Inability to cooperate with the scan process: inability to lie relatively still and in supine for 30-60 minutes or patient body habitus above scanner dimensions

Exclusion criteria for HEBIS scan:

* GFR < 30 ml/min/1.73m2
* < 2 weeks after antiviral eradication therapy for hepatitis C
* Bilirubine > 30 µmol/l
* Relative contra-indications (possibly affecting liver function): opiates, barbiturates, somatostatine, colestyramine, rifampicine, atropine

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Ten to fifteen patients with a single liver metastasis who will be treated with SBRT, will be included to assess functional imaging using HEBIS before and 3-4 months after their treatment (SBRT). Patients are included in a single institute , NKI-AvL, in consecutive or convenient order.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Dose-effect relationship between radiation dose and liver function by comparing the change in liver function before and after SBRT | This is measured at baseline, before treatment, and after 3-4 months after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arntz PJW, Deroose CM, Marcus C, Sturesson C, Panaro F, Erdmann J, Manevska N, Moadel R, de Geus-Oei LF, Bennink RJ. Joint EANM/SNMMI/IHPBA procedure guideline for [99mTc]Tc-mebrofenin hepatobiliary scintigraphy SPECT/CT in the quantitative assessment of the future liver remnant function. HPB (Oxford). 2023 Oct;25(10):1131-1144. doi: 10.1016/j.hpb.2023.06.001. Epub 2023 Jun 2. PMID 37394397